CLINICAL TRIAL: NCT02615418
Title: A Novel Non Invasive Brain Stimulation,tDCS Based Treatment for Chronic Low Back Pain (CLBP)-Sourasky Medical Center-Tel Aviv
Brief Title: Non Invasive Brain Stimulation Treatment for CLBP
Acronym: NIBSTCLBP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NIBS NeuroScience Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NIBS-Sour-1
Record Dates: First submitted 2015-11-23; First posted 2015-11-26 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Chronic Low Back Pain (CLBP)
MeSH Terms: interventions — Physical Examination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fully active treatement (Active Comparator)
  Interventions: Device: NIBS system for evaluation and treatment utilizing non invasive brain stimulation
- partially active (Sham Comparator): first 2.5 weeks will receive sham treatment followed by active
  Interventions: Device: NIBS system for evaluation and treatment utilizing non invasive brain stimulation

INTERVENTIONS:
Device: NIBS system for evaluation and treatment utilizing non invasive brain stimulation

SUMMARY:
This trial is designed to preliminary evaluate the efficacy and safety of NIBS system for treatment of chronic low back pain (CLBP) (over 6 months). The trial is of a double blind sham controlled partial crossover design and will involve 2 weekly treatments and evaluations for 6 weeks, with 6 weeks follow-up. The goal of the study is to 1. Asses the CLBP change immediate and long term effect for the trial duration and follow-up. 2. Asses quality of life improvement as measure by sleep quality and questioners. 3. Asses long term neuronal changes or lack thereof in treated and untreated subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80
* CLBP as defined by the European guidelines.
* low back pain first week average NPRS>4.

Exclusion Criteria:

1. Acute low back pain (duration of less than 6 months) first week average NPRS> 4
2. Neurological illness causing structural brain damage (e.g. Stroke, TIA)
3. Psychiatric disease other than mood disorders
4. Current chronic use of medications with pro-epileptic properties
5. Known alcohol dependency
6. Use of alcohol within the previous 24 hours
7. History of loss of consciousness
8. Epilepsy or epilepsy in a first degree relative
9. Medical implants
10. Pregnancy
11. Illicit drug use or within the previous month

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Change in CLBP on a 0-10 Numerical Pain Rating Scale (NPRS) | Baseline to week 6 .

SECONDARY OUTCOMES:
Change From Baseline in Sleep Quality (0-10 Numerical Rating Scale Scores) | Baseline to 6 weeks
Change CLBP quality of life -Roland-Morris questionnaire | Baseline to 6 weeks